CLINICAL TRIAL: NCT00904189
Title: Measurement of the Radiation Dose Cuticles Using Electron Paramagnetic Resonance (EPR) Spectroscopy
Brief Title: Measurement of the Radiation Dose Cuticles Using Electron Paramagnetic Resonance (EPR)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has relocated
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: U4706; RSRB00014685 (Other: University of Rochester IRB)
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Irradiation; Adverse Effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standard of care radiation therapy (No Intervention): Standard of care given for treatment of cancer. Subjects receiving incidental radiation dose to fingernails.
  Interventions: Radiation: Standard of care given for treatment of cancer

INTERVENTIONS:
Radiation: Standard of care given for treatment of cancer — Subjects receiving a known dose of radiation during Total Body Irradiation.

SUMMARY:
This study is to test the effectiveness a new method (called EPR dosimetry) that could be used to measure radiation doses to fingernails that occur as a result of unplanned exposure to radiation, such as might occur from the actions of terrorists, or from accidents.

DETAILED DESCRIPTION:
In the event of a radiological exposure incident, such as the detonation of a radiological dispersion device (RDD) in a terrorist attack or accidental exposures to sources of ionizing radiation, it is advantageous to use multiple methods to assess the dosimetry of individuals exposed to this radiation (4). These methods should include a physical assessment of the dosimetry at the exposure site to, 1) identify the type of radiation (e.g., gamma rays, neutrons or radioisotopes), 2) evaluate the distribution of radioisotopes and/or radioactivity at the site, and 3) determine the location of exposed individuals to the source of radiation. For individuals affected by the radiological incident, the monitoring of their clinical signs and symptoms is important for determining whether acute symptoms of radiation sickness are being presented and if immediate medical intervention is required. However, it is recognized that an invaluable aid for the clinical management of exposed individuals is the use of biomarkers that can be readily obtained from the exposed individual and used for assessing dosimetry (4,9). Biomarkers that are most useful to the physician are those produced or expressed within minutes to hours following exposure. With the dosimetry provided through these early phase biomarker measurements, the physician can better assess the clinical signs that are presented by an exposed individual and better determine the need and course of treatment.

ELIGIBILITY:
Inclusion Criteria:

Arm 1:

* Radiation field to include one or more fingernail or toenail;
* KPS > 70;
* For TBI subjects: sufficient cuticle length (3 mm or greater) on all fingers and/or toes.

Exclusion Criteria:

* Prior therapeutic radiation doses to the fingernails;
* Life expectancy < 6 months;
* lifetime radiation dose of greater than 0.1 Gy through prior radiation therapy or occupational exposures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Swarts, PhD, Principal Investigator — Department of Radiation Oncology, University of Rochester Medical Center
Locations (1):
- Department of Radiation Oncology, University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Subjects Receiving Incidental Radiation Dose to Fingernails.: Subjects receiving incidental radiation dose to fingernails.
  Standard of care given for treatment of cancer: Subjects receiving a known dose of radiation during Total Body Irradiation.
Period: Overall Study
Arm/Group | 1 Subjects Receiving Incidental Radiation Dose to Fingernails.
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 1Subjects Receiving Incidental Radiation Dose to Fingernails.: Subjects receiving incidental radiation dose to fingernails.
  Standard of care given for treatment of cancer: Subjects receiving a known dose of radiation during Total Body Irradiation.
Arm/Group | 1Subjects Receiving Incidental Radiation Dose to Fingernails.
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Dose of Radiation Received by Fingernails
Description: The mean dose in gray of radiation exposure to participants fingernails as determined by Electron Paramagnetic Resonance (EPR).
Time Frame: 2.5 years
Population: The study enrolled only 2 subjects and then was substantially changed. After the amendment, no further subjects were enrolled. The data collected from the two enrolled subjects was not analyzed and therefore is not available.
Groups:
- Subjects Receiving Incidental Radiation Dose to Fingernails.: Subjects receiving incidental radiation dose to fingernails.
  Standard of care given for treatment of cancer: Subjects receiving a known dose of radiation during Total Body Irradiation.
Arm/Group | Subjects Receiving Incidental Radiation Dose to Fingernails.
Number analyzed (Participants) | 0

2. Secondary Outcome: Determination of the Range of Background Signal Measured by the EPR Device.
Time Frame: 2.5 years
Population: as for outcome 1
Arm/Group | 1 Subjects Receiving Incidental Radiation Dose to Fingernails.
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Subjects Receiving Incidental Radiation Dose to Fingernails.
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes